CLINICAL TRIAL: NCT00971022
Title: Discount Generic Prescription Utilization in Low-income Populations
Brief Title: Discount Generic Prescription Study
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0340
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Poverty; Low-Income Population
Keywords: Low-income populations; Chronic health condition; Prescription medication; Prescription drugs; Discount generic prescription programs; Survey; Awareness; Focus Group; Houston
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low-income Populations
  Interventions: Behavioral: Survey; Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Survey — 20 minute survey to determine the relationship between awareness of the discount generic prescription program and utilization of the program.
  Other Names: Questionnaire
Behavioral: Focus Group — 5 - 8 focus groups of 6 - 10 people, lasting approximately 90 minutes

SUMMARY:
The goal of this study is to learn about the factors that influence people to take part in discount generic prescription programs.

The primary objective of this study is to identify the factors associated with awareness and utilization of discount generic prescription programs and how two low-income populations in Houston utilize the $4 for a 30-day supply or $10 for a 90-day supply, Generic Prescriptions Program offered by Kroger, Randalls, Target, Walmart, HEB, CVS, and Walgreens.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will take part in a focus group. The focus group will consist of about 8 people who will discuss beliefs about generic medication, awareness of discount generic prescription programs, and use of the discount generic prescription program. The focus group will last about 90 minutes.

During the focus group, you will complete a form that asks for basic demographic information (such as your age and sex).

The focus group discussions will be taped, and the recorded tapes will be transcribed word-for-word. The taped recording of the focus group study will be stored in a safe and secured locker by the study chair. The taped recordings will be destroyed after 5 years.

Length of Study:

Your participation on this study will end once you complete the focus group.

This is an investigational study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Low-income (less than $30,000/year)
* Ability to speak English
* Ability to read and write in English
* Chronic health condition requiring prescription medication or family member with chronic health condition requiring prescription medication.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults or an adult's family member, over the age of 18, with a low-income (less than $30,000/year) and a chronic health condition requiring prescriptions.
Sampling Method: Non-Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of low-income adults who are aware of discount generic prescription programs (Survey) | 12 Months (estimated survey completion time 20 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Lovell A. Jones, PHD, BS, MA, Study Chair — UT MD Anderson Cancer Center; Anthony Omojasola, DRPH, Principal Investigator — UT MD Anderson Cancer Center
Locations (3):
- United States (3):
  - Independence Heights Community Health Center, Houston, Texas
  - HOPE Clinic, Houston, Texas
  - Second Mile Mission Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org